CLINICAL TRIAL: NCT01462201
Title: A Multicenter,Two-Arm,Randomized,Controlled Study for the Evaluation of the Treatment of Adipose Tissue Using a Focused Ultrasound Device
Brief Title: A Multicenter,2-Arm,Randomized,Controlled Study Evaluate the Effectiveness of the UltraShape® Contour I VER 3.1 System for Non-Invasive Reduction in Abdominal Circumference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UltraShape (Industry)
Collaborators: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: US-0711
Record Dates: First submitted 2011-10-17; First posted 2011-10-31 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Body Sculpting
Keywords: focused ultrasound; mechanical fat destruction; Body Sculpting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - Non Invasive Ultrasound (Experimental): Group 1 3 visits - Measurement of abdominal circumferences 3 visits - Treatment with Ultrashape Contour I VER 3.1 4 visits - Follow up visits The intervention is non invasive ultrasound.
  Interventions: Device: Non Invasive Ultrasound
- Group 2 - Non Invasive Ultrasound (Experimental): Group 2 3 visits - Treatment with Contour I VER 3.1 system 3 visits - Measurements of abdominal circumference 4 visits - Follow Up visits The intervention is non invasive ultrasound.
  Interventions: Device: Non Invasive Ultrasound

INTERVENTIONS:
Device: Non Invasive Ultrasound — Each treatment session is estimated to take approximately 60 minutes and will be performed on a bi-weekly basis.

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of the Contour I VER 3.1 System on abdominal midsection circumference reduction relative to no treatment.

The secondary objective of this study is to assess subject satisfaction measured with a self-assessment questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subjects, 18 and 65 years of age at the time of enrollment
2. Abdominal fat thickness of at least 1.5 cm (measurement by caliper)
3. For women of child-bearing potential:

   1. negative urine pregnancy test.
   2. Women of child bearing age are required to be using an acceptable form of birth control for the duration of the study.
4. General good health confirmed by medical history and skin examination of the treated area
5. Written informed consent to participate in the study
6. Ability to comply with the requirements of the study
7. BMI ≤ 30

   Intra-procedural Inclusion criteria (prior to starting the treatment phase):

   subjects are eligible to continue the study and participate in the treatment phase if she meets all of the following intra-procedural inclusion criteria:
8. For women of child-bearing potential: negative pregnancy test
9. Abdominal fat thickness of at least 1.5 cm prior to initial treatment (measurement by caliper)

Exclusion Criteria:

1. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker/defibrillator, abdominal aortic aneurysm
2. Current hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease or malignancy.
3. Previous liposuction in the treatment area
4. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing
5. Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions) including depressed scars in the treatment area
6. Poor skin quality (i.e., laxity)
7. Abdominal wall diastasis or hernia on physical examination
8. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months
9. Obesity (BMI > 30)
10. Childbirth within the last 12 months or breastfeeding women.
11. Any acute or chronic condition which, in the opinion of the Investigator, could interfere with the conduct of the study
12. Unstable weight within the last 6 months (i.e., ± 3% weight change in the prior six months)
13. Inability to comply with circumference measurement procedure (e.g., inability to held breath for the required duration)
14. Participation in another clinical study within the last six months.
15. Previous body contouring treatments in the areas of the abdomen and flanks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the effectiveness of the Contour I VER 3.1 System on abdominal midsection circumference reduction relative to no treatment | 5-6 months
  Reduction in circumference measurement of the abdomen from baseline

SECONDARY OUTCOMES:
Assess subject satisfaction measured with a self-assessment questionnaire | 5-6 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Dr. William Patrick Coleman, III, Metairie, Louisiana
  - MD Laser Skin & Vein Institute, Hunt Valley, Maryland
  - New-Jersey Plastic Surgery, Montclair, New Jersey
  - Dr. Jeffrey Kenkel, Dallas, Texas
- Department of Plastic Surgery and Burns Rabin Medical Center - Beilinson Hospital, Petah Tikva, Israel